CLINICAL TRIAL: NCT00716482
Title: Assessment of the Clinical Value of SuperSonic Shear Wave Elastography in the Ultrasonic Evaluation of Breast Lesions
Brief Title: Ultrasound Elastography of Breast Lesions
Acronym: BE1
Status: Completed | Type: Observational
Sponsor: SuperSonic Imagine (Industry)
Responsible Party: Sponsor
Other Study IDs: A00152-53
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Results first posted 2013-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Breast Neoplasms
Keywords: breast; lesion; ultrasound; BI-RADS; malignancy; women
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Our hypothesis is that the addition of ShearWave Elastography (SWE) to a conventional breast ultrasound examination provides useful information for the radiologist when imaging lesions in the breast, as compared to conventional grayscale ultrasound alone.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been referred to a breast ultrasound because of a positive physical palpation and/or positive mammograms and/or positive ultrasound and/or positive MRI.
* female
* age 21 or older
* provide informed consent

Exclusion Criteria:

* Women who are unwilling or unable to provide informed consent
* Women with breast implants
* Women with superficial lesions or lesions on skin (with the most superficial surface of the lesion within 5 mm of the skin surface)
* Women who are pregnant or breastfeeding
* Women who are undergoing chemotherapy or radiotherapy for any cancer
* Women with previous breast conserving surgery on the breast of interest Note: Previous excision of a benign lesion 4 cm or more away from the suspected lesion does not constitute an exclusion criterion.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will consist of women who have been referred to a public or private hospital or clinic for a breast ultrasound evaluation. The sites are located various cities throughout the United States and Europe.
Sampling Method: Non-Probability Sample
Enrollment: 1681 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O Cosgrove, MD, Principal Investigator — Hammersmith Hospitals NHS Trust
Locations (16):
- United States (6):
  - University of Southern California - LAC+USC Medical Center, OPD Rm 3P61, Los Angeles, California
  - Sally Jobe Breast Center, Denver, Colorado
  - Yale Medical Center, Department of Diagnostic Radiology, New Haven, Connecticut
  - Northwestern Memorial Hospital, Dept. of Radiology, Chicago, Illinois
  - Boston Medical Center, Radiology, Boston, Massachusetts
  - Thomas Jefferson Medical Center, Department of Radiology, Philadelphia, Pennsylvania
- France (4):
  - Hôpital Privé Jean Mermoz, Lyon
  - University Hospital La Timone, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
- Germany (4):
  - University Hospital, Frauenklinik, Greifswald
  - University Hospital Schleswig-Holstein, Kiel
  - Marienhospital, Klinik für Radiologie, Osnabrück
  - German Diagnostic Clinic, Wiesbaden
- Ospedale Civile di Gorizia, Gorizia, Italy
- Charings Cross Hospital, London, United Kingdom

REFERENCES:
- [Result] Cosgrove DO, Berg WA, Dore CJ, Skyba DM, Henry JP, Gay J, Cohen-Bacrie C; BE1 Study Group. Shear wave elastography for breast masses is highly reproducible. Eur Radiol. 2012 May;22(5):1023-32. doi: 10.1007/s00330-011-2340-y. Epub 2011 Dec 31. PMID 22210408
- [Result] Berg WA, Cosgrove DO, Dore CJ, Schafer FK, Svensson WE, Hooley RJ, Ohlinger R, Mendelson EB, Balu-Maestro C, Locatelli M, Tourasse C, Cavanaugh BC, Juhan V, Stavros AT, Tardivon A, Gay J, Henry JP, Cohen-Bacrie C; BE1 Investigators. Shear-wave elastography improves the specificity of breast US: the BE1 multinational study of 939 masses. Radiology. 2012 Feb;262(2):435-49. doi: 10.1148/radiol.11110640. PMID 22282182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: October 23, 2008 - June 15, 2010 Hospitals and private medical clinics in 16 sites worldwide participated.
Groups:
- Breast Lesion: B-mode ultrasound examination with currently marketed machine followed by ultrasound B-mode examination and ShearWave Elastography examination
Period: Overall Study
Arm/Group | Breast Lesion
Started | 1681
Completed | 1562
Not Completed | 119
Not completed — Lost to Follow-up | 6
Not completed — Inadequate acquisition or analysis | 50
Not completed — no pathology obtained | 10
Not completed — technical/machine error | 28
Not completed — inclusion/exclusion criteria not met | 25

BASELINE CHARACTERISTICS:
Population: There were 1681 "started" participants and 1562 "completed" participants. Reasons for rejected participants are listed in "participant flow" section
Arm/Group | Breast Lesion
Number analyzed (Participants) | 1681
Age Continuous [Mean (Standard Deviation); unit: years] — mean age is based on 1681 participants
  years | 51.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1681
  Male | 0
Region of Enrollment [Number; unit: participants]
  France | 322
  United States | 566
  Germany | 529
  Italy | 89
  United Kingdom | 175

OUTCOME MEASURES:

1. Primary Outcome: Estimates of Effect of Selectively Upgrading BIRADS Category 3 and Downgrading BIRADS 4a Masses Based on SWE Features. Overall Specificity and Sensitivity of BI-RADS Score Using Conventional B-mode Ultrasound vs. B-mode + Certain SWE Characteristics
Description: Positive reference standard = malignant cytologic or histopathologic result. Negative reference standard = BIRADS 2 lesions, BIRADS 3 lesions with benign histopathology, or a 1 year follow-up ultrasound exam showing resolved or decreased lesion size.
  Conservative strategy:features of E-homogeneity, E-max and E-color were used to upgrade BIRADS 3 lesions to BIRADS 4a' or downgrade BIRADS 4a lesions to BIRADS 3'. Aggressive strategy used the same features but upgraded and downgraded more lesions.
  Based on 939 lesions.
Time Frame: 2 years
Population: Per protocol. Analysis includes 289 malignant and 650 benign masses. One lesion was analyzed per participant.
Measure: Number; unit: participants
Groups:
- Specificity: Number of benign lesions with negative test results/total number of benign lesions B-mode ultrasound examination with currently marketed machine followed by ultrasound B-mode examination and ShearWave Elastography examination
- Sensitivity: Number of cancers with positive test results/total #number of cancers B-mode ultrasound examination with currently marketed machine followed by ultrasound B-mode examination and ShearWave Elastography examination
Arm/Group | Specificity | Sensitivity
Number analyzed (Participants) | 650 | 289
participants
  lesion shape | 451 | 283
  lesion homogeneity-conservative strategy | 464 | 280
  lesion homogeneity-aggressive strategy | 510 | 278
  maximum elasticity (Emax)-conservative strategy | 427 | 286
  maximum elasticity (Emax)-aggressive strategy | 503 | 281
  median mean elasticity (Emean) | 407 | 285
  diameter ration (Edia) | 333 | 286
  median elasticity ratio (Erat) | 422 | 284
  color score of Emax (Ecol)-conservative strategy | 457 | 288
  color score of Emax (Ecol)-aggressive strategy | 510 | 285
Statistical Analysis 1: Comparison: Specificity; Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p < 0.001, McNemar — P-value was that to test the null hypothesis that there is no change in specificity with addition of the ShearWave elastographic feature. Significance threshold P-value = 0.05; Specificity of lesion shape = 0.694
Statistical Analysis 2: Comparison: Specificity; Elastography image specificity of the homogeneity of elasticity with the lesion and surrounding tissue using conservative strategy (BIRADS 3 mass upgraded to BIRADS 4a' if they were not homogeneous on the color overlay SW elastographic image; BIRADS 4a mass downgraded to BIRADS 3' if they were very homogeneous). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p < 0.001, McNemar — [p-value comment as in outcome 1, analysis 1]; Lesion homogeneity spec, conservative = 0.714
Statistical Analysis 3: Comparison: Specificity; Elastography image specificity of the homogeneity of elasticity with the lesion and surrounding tissue using aggressive strategy (BIRADS 3 mass upgraded to BIRADS 4a' if they were not homogeneous on the color overlay SW elastographic image; BIRADS 4a mass downgraded to BIRADS 3' if they were very or reasonably homogeneous). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p < 0.001, McNemar — [p-value comment as in outcome 1, analysis 1]; Lesion homogeneity spec, agressive = 0.785
Statistical Analysis 4: Comparison: Specificity; Elastography image specificity of the maximum elasticity using conservative strategy (BIRADS 3 mass upgraded to BIRADS 4a' if maximum elasticity was 160 kiloPascals (kPa) (7.3 m/sec) or more; BIRADS 4a mass downgraded to BIRADS 3' if the maximum elasticity was 30 kPa (3.2 m/sec) or less). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.001, McNemar — [p-value comment as in outcome 1, analysis 1]; Max. elasticity specificity,conservative = 0.657
Statistical Analysis 5: Comparison: Specificity; Elastography image specificity of the maximum elasticity using aggressive strategy (BIRADS 3 mass upgraded to BIRADS 4a' if maximum elasticity was 160 kPa(7.3 m/sec) or more; BIRADS 4a mass downgraded to BIRADS 3' if the maximum elasticity was 80 kPa (5.2 m/sec) or less). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p < 0.001, McNemar — [p-value comment as in outcome 1, analysis 1]; Max. elasticity specificity, aggressive = 0.774
Statistical Analysis 6: Comparison: Specificity; Elastography image median mean elasticity value. Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.18, McNemar — [p-value comment as in outcome 1, analysis 1]; median mean elasticity value specificity = 0.626
Statistical Analysis 7: Comparison: Specificity; Elastography image diameter ratio. Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.006, McNemar — [p-value comment as in outcome 1, analysis 1]; Diameter ratio specificity = 0.512
Statistical Analysis 8: Comparison: Specificity; Elastography image median elasticity ratio. Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.006, McNemar — [p-value comment as in outcome 1, analysis 1]; Median elasticity ratio specificity = 0.649
Statistical Analysis 9: Comparison: Specificity; Elastography image specificity of color using a six-point color scale of maximum elasticity in the mass and surrounding parenchyma using conservative strategy (BIRADS 3 mass upgraded to BIRADS 4a' if the max stiffness on the color overlay SW elastographic image was red; BIRADS 4a mass downgraded to BIRADS 3' if the max stiffness on the color overlay SW elastographic image was black to dark blue). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p < 0.001, McNemar — [p-value comment as in outcome 1, analysis 1]; Max.color scale specificity,conservative = 0.703
Statistical Analysis 10: Comparison: Specificity; Elastography image specificity of color using a six-point color scale of maximum elasticity in the mass and surrounding parenchyma using aggressive strategy (BIRADS 3 mass upgraded to BIRADS 4a' if the max stiffness on the color overlay SW elastographic image was red; BIRADS 4a mass downgraded to BIRADS 3' if the max stiffness on the color overlay SW elastographic image was black to dark blue, or light blue). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p < 0.001, McNemar — P-value was that to test the null hypothesis that there is no change in specificity with addition of the ShearWave elastographic feature. Significance threshold P-value = 0.05 Overall specificity = 78.5%; Max. color scale specificity, aggressive = 0.785
Statistical Analysis 11: Comparison: Sensitivity; Elastography image lesion shape. Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.48, McNemar — P-value was that to test the null hypothesis that there is no change in sensitivity with addition of the ShearWave elastographic feature. Significance threshold P-value = 0.05; Lesion shape sensitivity = 0.979
Statistical Analysis 12: Comparison: Sensitivity; Elastography image sensitivity of the homogeneity of elasticity with the lesion and surrounding tissue using conservative strategy (BIRADS 3 mass upgraded to BIRADS 4a' if they were not homogeneous on the color overlay SW elastographic image; BIRADS 4a mass downgraded to BIRADS 3' if they were very homogeneous). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.74, McNemar — [p-value comment as in outcome 1, analysis 11]; Lesion homogeneity sens, conservative = 0.969
Statistical Analysis 13: Comparison: Sensitivity; Elastography image sensitivity of the homogeneity of elasticity with the lesion and surrounding tissue using aggressive strategy (BIRADS 3 mass upgraded to BIRADS 4a' if they were not homogeneous on the color overlay SW elastographic image; BIRADS 4a mass downgraded to BIRADS 3' if they were very or reasonably homogeneous). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.37, McNemar — [p-value comment as in outcome 1, analysis 11]; elasticity homogeneity,aggressive,sensit = 0.962
Statistical Analysis 14: Comparison: Sensitivity; Elastography image sensitivity of the maximum elasticity using conservative strategy (BIRADS 3 mass upgraded to BIRADS 4a' if maximum elasticity was 160 kPa(7.3 m/sec) or more; BIRADS 4a mass downgraded to BIRADS 3' if the maximum elasticity was 30 kPa (3.2 m/sec) or less). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.025, McNemar — P-value was that to test the null hypothesis that there is no change in sensitivity with addition of the ShearWave elastographic feature. Significance threshold P-value = 0.05 Overall sensitivity = 99.0%; elasticity homegeneity,conservative,sens = 0.990
Statistical Analysis 15: Comparison: Sensitivity; Elastography image sensitivity of the maximum elasticity using aggressive strategy (BIRADS 3 mass upgraded to BIRADS 4a' if maximum elasticity was 160 kPa(7.3 m/sec) or more; BIRADS 4a mass downgraded to BIRADS 3' if the maximum elasticity was 80 kPa (5.2 m/sec) or less). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p > 0.99, McNemar — [p-value comment as in outcome 1, analysis 11]; max. elasticity sensitivity,aggressive = 0.972
Statistical Analysis 16: Comparison: Sensitivity; Elastography image median mean elasticity value. Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.046, McNemar — [p-value comment as in outcome 1, analysis 11]; median mean elasticity value sensitivity = 0.986
Statistical Analysis 17: Comparison: Sensitivity; Elastography image diameter ratio. Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.025, McNemar — [p-value comment as in outcome 1, analysis 11]; diameter ratio sensitivity = 0.990
Statistical Analysis 18: Comparison: Sensitivity; Elastography image median elasticity ratio. Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.083, McNemar — [p-value comment as in outcome 1, analysis 11]; median elasticity ratio sensitivity = 0.983
Statistical Analysis 19: Comparison: Sensitivity; Elastography image sensitivity of color using a six-point color scale of maximum elasticity in the mass and surrounding parenchyma using conservative strategy (BIRADS 3 mass upgraded to BIRADS 4a' if the max stiffness on the color overlay SW elastographic image was red; BIRADS 4a mass downgraded to BIRADS 3' if the max stiffness on the color overlay SW elastographic image was black to dark blue). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.008, McNemar — [p-value comment as in outcome 1, analysis 11]; Max.color scale sensitivity,conservative = 0.997
Statistical Analysis 20: Comparison: Sensitivity; Elastography image sensitivity of color using a six-point color scale of maximum elasticity in the mass and surrounding parenchyma using aggressive strategy (BIRADS 3 mass upgraded to BIRADS 4a' if the max stiffness on the color overlay SW elastographic image was red; BIRADS 4a mass downgraded to BIRADS 3' if the max stiffness on the color overlay SW elastographic image was black to dark blue, or light blue). Null hypothesis is that there is no difference between the two tests; Test type: Superiority or Other; p = 0.21, McNemar — [p-value comment as in outcome 1, analysis 11]; Max. color scale sensitivity, aggressive = 0.986

2. Secondary Outcome: Qualitative Intraobserver Reproducibility of SWE Related to Homogeneity Feature
Description: 614 benign and 144 malignant breast lesions were scanned in SWE 3 consecutive times, and the similarity of the 3 images was evaluated by the investigator.
Time Frame: performed on the same day, within 2 years from study start date
Population: Per protocol. One lesion was analyzed per participant.
Measure: Number; unit: participants
Groups:
- Very Homogeneous: The Elastography image of the lesion has a smooth and consistent color appearance throughout, or very subtle color differences relating to small changes on the color scale are observed.
- Reasonably Homogeneous: The Elastography image of the lesion has a slightly "patchy" appearance. The image may consist of larger (2-5mm) sub-regions within the lesion boundary that are homogenous, or the color differences between adjacent areas within the lesion are small.
- Not Homogeneous: The Elastography image of the lesion is inhomogeneous and has a "mottled" or "patchy" appearance throughout.
Arm/Group | Very Homogeneous | Reasonably Homogeneous | Not Homogeneous
Number analyzed (Participants) | 391 | 212 | 155
participants
  All images very or reasonably similar | 385 | 176 | 105
  Some images similar | 5 | 34 | 45
  Images very dissimilar | 1 | 2 | 5
Statistical Analysis 1: Comparison: Very Homogeneous vs Reasonably Homogeneous vs Not Homogeneous; Null hypothesis: no variance of similarity exists between the three groups; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis; Kruskal-Wallis one-way ANOVA. Kruskal-Wallis was performed once to get p-values for all of the 9 categories at once

3. Secondary Outcome: Intraobserver Reliability of Quantitative SWE Measurements
Description: 614 benign and 144 malignant lesions. Each category's measurement (diameter, area, etc..) is performed 3 times. These 3 measurements are then compared with each other in order to calculate the interclass correlation coefficient.
Time Frame: performed on the same day, within 2 years from study start date
Population: Per protocol. 758 masses (614 benign and 144 malignant)are analyzed. One lesion was analyzed per participant. 3 acquisitions per lesion were analyzed with the ICC method for 10 different parameters.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- Overall (All Masses): 614 benign and 144 malignant masses
Arm/Group | Overall (All Masses)
Number analyzed (Participants) | 758
correlation coefficient
  Diameter | 0.94 [0.94 to 0.95]
  Area | 0.95 [0.94 to 0.95]
  Perimeter | 0.95 [0.94 to 0.95]
  E minimum mass | 0.71 [0.68 to 0.74]
  E maximum mass | 0.84 [0.82 to 0.86]
  E mean mass | 0.87 [0.85 to 0.88]
  E ratio (mass:fat) | 0.77 [0.74 to 0.79]
  E minumum fat | 0.57 [0.53 to 0.61]
  E maximum fat | 0.62 [0.58 to 0.65]
  E mean fat | 0.71 [0.68 to 0.74]

4. Secondary Outcome: Interobserver Agreement of B Mode Ultrasound and SWE Features
Description: 614 benign and 144 malignant breast masses.
Time Frame: performed on the same day, after study completion
Population: Per protocol. One lesion was analyzed per participant. Two independent readers did a qualitative assessment of 7 image parameters (per lesion) using Kappa.
Measure: Number (95% Confidence Interval); unit: kappa statistic
Groups:
- Overall (All Masses): Benign and malignant lesions
Arm/Group | Overall (All Masses)
Number analyzed (Participants) | 758
kappa statistic
  B-mode shape | 0.58 [0.51 to 0.65]
  B-mode orientation | 0.53 [0.46 to 0.60]
  B-mode margin | 0.38 [0.32 to 0.45]
  B-mode BI-RADS assessment | 0.59 [0.53 to 0.66]
  SWE shape | 0.40 [0.33 to 0.47]
  SWE homogeneity | 0.57 [0.51 to 0.64]
  SWE Emax | 0.66 [0.59 to 0.73]

ADVERSE EVENTS:
Description: Adverse Events were not collected as a part of this study.
Arm/Group | Breast Lesion
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
* follow up on BI-RADS 2 lesions was not performed
* operators knew the BI-RADS score of the lesion before performing SWE
* more BI-RADS 3 and 4 lesions were recruited because of the study design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No